CLINICAL TRIAL: NCT02170714
Title: Managing Pediatric Acute Severe Colitis According to the 2011 ECCO-ESPGHAN Guidelines: Efficacy of Infliximab as a Rescue Therapy
Brief Title: Efficacy of Infliximab as a Rescue Therapy in Pediatric Acute Severe Colitis
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Marina Aloi, Assistant Professor, University of Roma La Sapienza
Other Study IDs: 16062014
Record Dates: First submitted 2014-06-16; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Pediatric Acute Severe Colitis
Keywords: Acute severe colitis; Children; Infliximab; colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ASC: Consecutive children hospitalized for an episode of acute ASC, defined as a PUCAI > 65. All patients were treated according to the 2011 ECCO-ESPGHAN guidelines for ASC: all patients received intravenous (iv) corticosteroids (methylprednisolone 1.5-2 mg/Kg/day) for 5 days. Patients not responding to corticosteroids (i.e. PUCAI>65 at day 5) started Infliximab (IFX, 5 mg/Kg 0,2,6 then every 8 weeks) as second-line therapy. All therapies were decided at the discretion of the referral gastroenterologist and recorded on standardized case report forms. A follow-up of 2 years for the colectomy risk was evaluated for all patients.
  Interventions: Other: Clinical and laboratory assessment

INTERVENTIONS:
Other: Clinical and laboratory assessment — Clinical assessment through PUCAI and laboratory data (Erythrocyte Sedimentation Rate, C-Reactive Protein, hemoglobin, albumin, hematocrit, ferritin) were recorded at admission and at day 3 and 5. All patients were treated according to the 2011 ECCO-ESPGHAN guidelines for ASC: all patients received intravenous (iv) corticosteroids (methylprednisolone 1.5-2 mg/Kg/day) for 5 days. Patients not responding to corticosteroids (i.e. PUCAI>65 at day 5) started Infliximab (IFX, 5 mg/Kg 0,2,6 then every 8 weeks) as second-line therapy. All therapies were decided at the discretion of the referral gastroenterologist and recorded on standardized case report forms

SUMMARY:
Background and aims: Acute severe ulcerative colitis (ASC) is a potentially life-threatening event. Poor pediatric data are available about the success rates of Infliximab (IFX) as a second line therapy. This study was performed in consecutively observed pediatric patients with ASC, treated according to the 2011 European Crohn's colitis Organization (ECCO)- European Society for Pediatric Gastroenterology, Hepatology and nutrition (ESPGHAN) guidelines on pediatric ASC¹ and aim to assess the long-term efficacy of IFX and clinical predictors of poor outcome.

Methods: Children hospitalized for an episode of ASC, defined as a Pediatric Ulcerative Colitis Activity Index (PUCAI) of at least 65 points, were enrolled. Clinical assessment through PUCAI and laboratory data (Erythrocyte Sedimentation Rate, C-Reactive Protein, hemoglobin, albumin, hematocrit, ferritin) was recorded at admission and at day 3 and 5. All patients were treated according to the above mentioned guidelines for ASC and received intravenous (iv) corticosteroids (CS) as first-line therapy. IFX was administered as second-line therapy in CS-refractory patients. In a 2-year follow up the overall colectomy rate and the efficacy of IFX in avoiding colectomy were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ASC
* Confirmed diagnosis of ulcerative colitis (UC)
* Age 1-18 years

Exclusion Criteria:

* Not confirmed diagnosis of UC
* Contraindications for infliximab therapy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Consecutive children hospitalized for an episode of ASC, defined as a PUCAI>65
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The number of patients with ASC treated with IFX requiring colectomy | 24 months
  The surgical need will be evaluated in the group of patients treated with IFX during a 24-month follow-up

SECONDARY OUTCOMES:
The number of patients with ASC requiring colectomy | 1,6,12,18,24 months
To identify clinical predictive factors at the diagnosis of ASC of surgical need at follow-up | First day of the hospitalization
  Clinical variables at the diagnosis of ASC (i.e. duration of the disease before the episode of SC, past and ongoing therapies, age, family history, Perinuclear Anti-Neutrophil Cytoplasmic Antibodies - pANCA, PUCAI) were evaluated in the group of children needed colectomy at follow-up versus those not requiring surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Background] Turner D, Travis SP, Griffiths AM, Ruemmele FM, Levine A, Benchimol EI, Dubinsky M, Alex G, Baldassano RN, Langer JC, Shamberger R, Hyams JS, Cucchiara S, Bousvaros A, Escher JC, Markowitz J, Wilson DC, van Assche G, Russell RK; European Crohn's and Colitis Organization; Porto IBD Working Group, European Society of Pediatric Gastroenterology, Hepatology, and Nutrition. Consensus for managing acute severe ulcerative colitis in children: a systematic review and joint statement from ECCO, ESPGHAN, and the Porto IBD Working Group of ESPGHAN. Am J Gastroenterol. 2011 Apr;106(4):574-88. doi: 10.1038/ajg.2010.481. Epub 2011 Jan 11. PMID 21224839
- [Background] Turner D, Griffiths AM. Acute severe ulcerative colitis in children: a systematic review. Inflamm Bowel Dis. 2011 Jan;17(1):440-9. doi: 10.1002/ibd.21383. PMID 20645317
- [Background] Turner D, Mack D, Leleiko N, Walters TD, Uusoue K, Leach ST, Day AS, Crandall W, Silverberg MS, Markowitz J, Otley AR, Keljo D, Mamula P, Kugathasan S, Hyams J, Griffiths AM. Severe pediatric ulcerative colitis: a prospective multicenter study of outcomes and predictors of response. Gastroenterology. 2010 Jun;138(7):2282-91. doi: 10.1053/j.gastro.2010.02.047. Epub 2010 Feb 26. PMID 20193683